CLINICAL TRIAL: NCT07190794
Title: Evaluation of Endoscopic Sleeve Gastroplasty (ESG) as an Alternative Weight Loss Strategy for Patients With Obesity Discontinuing GLP-1 Receptor Agonists Due to Intolerance or Ineffectiveness: A Retrospective Study
Brief Title: RESCUE: Discontinuation of GLP-1
Status: Recruiting | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: E7234
Record Dates: First submitted 2025-09-17; First posted 2025-09-24 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obesity
Keywords: GLP-1; ESG; OverStitch
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- ESG Recipients: After discontinuing GLP-1 medication, this group elected to have an ESG procedure as a weight loss treatment.
  Interventions: Device: OverStitch™ or OverStitch NXT™
- Lifestyle Modification: After discontinuing GLP-1 medication, this group elected to participate in a structured lifestyle modification program.
  Interventions: Behavioral: Lifestyle Modification

INTERVENTIONS:
Device: OverStitch™ or OverStitch NXT™ — The OverStitch™ or OverStitch NXT™ Endoscopic Suturing System was used as part of each patient's ESG procedure within the routine clinical practice.
  Groups: ESG Recipients
Behavioral: Lifestyle Modification — Patients participated in a lifestyle modification program for weight loss management.
  Groups: Lifestyle Modification

SUMMARY:
This study is designed to compare weight loss outcomes and safety of ESG versus lifestyle modification in patients with obesity who discontinued GLP-1 therapy due to intolerance or suboptimal weight loss.

DETAILED DESCRIPTION:
This retrospective cohort study includes collection of data from medical records for consecutively treated patients undergoing treatment for weight loss following GLP-1 discontinuation. Weight loss treatment is either ESG with OverStitch™ OverStitch NXT™ or matched timeframe controls who participated in a lifestyle modification program for weight loss management.

Subjects will be enrolled in a 2:1 ratio (ESG: Lifestyle modification)

Patients are required to have the following visits for weight loss management:

* Completed initial consultation visit (baseline) prior to initiation of weight management program with documented GLP-1 history and reason for discontinuation
* Initiation of weight loss management between August 2021 and September 2024
* A minimum of two weight loss management visits, defined as performed by the physician that is managing the weight loss program and/or an affiliated weight loss specialist, completed at 1, 3, 6, or 9 months from the initiation of weight loss management
* Completed 1-year weight loss management visit (as defined above)

ELIGIBILITY:
Inclusion Criteria:

1. Adults (≥ 18 years)
2. BMI ≥30 kg/m² and ≤ 50 kg/m2
3. Discontinued GLP-1 therapy for weight loss (semaglutide and tirzepatide only) for intolerance or suboptimal weight loss (<5% TBWL after 3 months at maximally tolerated dose)
4. Initiation of weight loss management between August 2021 and September 2024
5. Completed 1-year follow-up for weight loss management (ESG and lifestyle modification or lifestyle modification alone) following initiation of weight loss treatment
6. Completed at least two interim visits for weight loss management from 1, 3, 6, through 9 months following initiation of weight loss treatment

Exclusion Criteria:

1. Missing data regarding GLP-1 treatment history, including weight before GLP-1 treatment and at discontinuation, and discontinuation reason
2. History of GLP-1 medication for a reason other than weight management
3. Had bariatric surgery or an endoscopic procedure for weight loss treatment other than ESG with OverStitch™ or OverStitch NXT™ within 1 year of starting weight loss management
4. Had an additional endoscopic treatment performed prior to or at the time of the ESG procedure that could influence weight loss results
5. Had another weight loss treatment during the 1-year follow-up reported during this study. Weight loss treatment includes but is not limited to appetite suppressants, anti-obesity medications, plastic surgery or body contouring procedures.
6. Pregnancy during the 1 year following initiation of weight loss management

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults over 18 years of age who were prescribed GLP-1 medication for weight loss and discontinued it due to intolerance of symptoms or suboptimal weight loss.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Percent total body weight loss (TBWL) at 1 year from baseline | 12 months
  The study will measure the percentage of total body weight loss for a period of one year from baseline.

SECONDARY OUTCOMES:
Change in body mass index (BMI) | 12 months
  The study will measure change in BMI for a period of one year from baseline.
Percentage of excess weight loss | 12 months
  The study will measure the percentage of excess weight loss for a period of one year from baseline.
Percentage of patients that achieved 5%, 10% and 15% total body weight loss | 12 months
  The study will measure the percentage of patients that achieved 5%, 10% and 15% total body weight loss in the one year from baseline.
Metabolic markers, if available | 12 months
  Metabolic markers include changes from baseline in the following items:
  1. HbA1c
  2. Fasting blood glucose
  3. Total cholesterol
  4. LDL
  5. HDL
  6. Triglycerides
  7. Blood pressure (systolic and diastolic blood pressure)
Visit compliance and impact to responder rate | 12 months
  Responders are defined as >= 10% TBWL. This analysis will analyze if responder rate improves with higher visit compliance (number of completed interactions with a provider for weight loss management).
Rate of procedure-related serious adverse events within 1-year post-ESG | 12 months
  The study will examine the rate of procedure-related serious adverse events within 1-year post-ESG.

CONTACTS AND LOCATIONS:
Overall Officials: Pichamol Jirapinyo, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (3):
- United States (3):
  - Bariendo, Miami, Florida
  - Brigham & Women's Hospital, Boston, Massachusetts
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No